CLINICAL TRIAL: NCT02650037
Title: Estudio de validación de la pulsioximetría Como método diagnóstico no Invasivo de Atelectasia Pulmonar y de la Efectividad de la Maniobra de Capacidad Vital Para la reversión de la Atelectasia Durante el Postoperatorio
Brief Title: The Air Test: A New Simple, Non-invasive Method to Diagnose Anesthesia-induced Atelectasis
Status: Completed | Type: Observational
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Responsible Party: Principal Investigator, Carlos Ferrando, MD, PhD, Fundación para la Investigación del Hospital Clínico de Valencia
Other Study IDs: AirTest
Record Dates: First submitted 2015-12-28; First posted 2016-01-08 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Patients With ASA Status I-III Scheduled for Elective Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Air Test — The Air Test simply consisted in breathing room air for 5 min on arrival into the postoperative anesthesia care unit while measuring peripheral oxygen saturation by Pulse oximetry

SUMMARY:
Anesthesia-induced atelectasis persist in the postoperative period but are not usually diagnosed because imaging techniques are required. The aim of the study is to determine whether the value of SpO2≤96 while breathing room air (0.21 FiO2) for 5 min, maneuver that we defined as the Air Test, was able to diagnose atelectasis in the postoperative period after a general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* Scheduled for elective surgery

Exclusion Criteria:

* age of <18 years
* pregnant women
* previous lung resection
* local-regional anesthesia
* cardio-thoracic anesthesia
* preoperative room air SpO2 less than 97%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study included all patients with ASA status I-III scheduled for elective surgery.
Sampling Method: Non-Probability Sample
Enrollment: 181 (Actual)
Dates: Start 2014-11; Primary Completion 2015-02 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Presence of postoperative atelectasis meassured by SpO2 levels and confirmed by computed tomography. | 35 minutes post-surgery
  After arrival to the post-surgery unit, patients received supplemental oxygen through a venturi mask with flow adjusted to approximate a FiO2 of 0.5 during the first 30 minutes. The SpO2 measure was made removing the oxygen mask and leaving the patients to breath room air for at least for 5 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesia and Critical Care; Hospital Clinico Universitario, Valencia, Valencia, Spain

REFERENCES:
- [Background] Hemmes SN, Serpa Neto A, Schultz MJ. Intraoperative ventilatory strategies to prevent postoperative pulmonary complications: a meta-analysis. Curr Opin Anaesthesiol. 2013 Apr;26(2):126-33. doi: 10.1097/ACO.0b013e32835e1242. PMID 23385321
- [Background] Magnusson L, Spahn DR. New concepts of atelectasis during general anaesthesia. Br J Anaesth. 2003 Jul;91(1):61-72. doi: 10.1093/bja/aeg085. No abstract available. PMID 12821566
- [Background] Hedenstierna G, Tokics L, Strandberg A, Lundquist H, Brismar B. Correlation of gas exchange impairment to development of atelectasis during anaesthesia and muscle paralysis. Acta Anaesthesiol Scand. 1986 Feb;30(2):183-91. doi: 10.1111/j.1399-6576.1986.tb02393.x. PMID 3085429
- [Derived] Ferrando C, Romero C, Tusman G, Suarez-Sipmann F, Canet J, Dosda R, Valls P, Villena A, Serralta F, Jurado A, Carrizo J, Navarro J, Parrilla C, Romero JE, Pozo N, Soro M, Villar J, Belda FJ. The accuracy of postoperative, non-invasive Air-Test to diagnose atelectasis in healthy patients after surgery: a prospective, diagnostic pilot study. BMJ Open. 2017 May 29;7(5):e015560. doi: 10.1136/bmjopen-2016-015560. PMID 28554935